CLINICAL TRIAL: NCT01289587
Title: Efficacy and Feasibility of a Program to Promote Physical Activity in Patients With Type 2 Diabetes (DIAfit)
Brief Title: Promoting Physical Activity in Patients With Type 2 Diabetes (DIAfit)
Acronym: DIAfit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Jardena Puder, MD, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 252/10
Record Dates: First submitted 2011-01-28; First posted 2011-02-04 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Diabetes
Keywords: Diabetes; Physical activity; Body composition; Aerobic fitness; Metabolic control
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alternative frequency variant (Experimental): An alternative variant of the DIAfit program (progressive increase of the number of administered PA sessions per week, namely one PA session per week during 4 weeks and then twice a week over a period of 16 weeks)
  Interventions: Behavioral: Physical activity intervention
- Standard frequency program (Active Comparator): Standard usual program (3 times per week over a period of 12 weeks)
  Interventions: Behavioral: Physical activity intervention

INTERVENTIONS:
Behavioral: Physical activity intervention — 36 sessions of physical activity offered at different frequencies

SUMMARY:
The aim of this study is to evaluate the effects of a physical activity intervention in patients with type 2 diabetes in a community setting.

DETAILED DESCRIPTION:
The aim of this study is

1. to evaluate the effects (before and after) of a physical activity program (DIAfit program) which contains 36 sessions of structured PA and also encourages unstructured PA in an unselected population of patients with type 2 diabetes independent of the selected variant of the program
2. to compare the effects of a standard DIAfit program (3 times per week for 12 weeks) with and alternative program which suggests a more progressive PA activity intensity (starting with one PA session per week during 4 weeks and then twice a week over a period of 16 more weeks (20 weeks total). In total the program also consist of 36 sessions)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes

Exclusion Criteria:

* Orthopedic complications
* Diabetic foot ulceration
* "Active " cardiac (ischemia during the exercise test) or stade III peripheral vascular disease
* Untreated proliferative retinopathy
* Autonomic neuropathy
* Active psychiatric, neurological, orthopedic, muscular or rheumatic disease interfering with a participation in a physical activity program
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2011-02; Primary Completion 2012-12 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Aerobic fitness | End of the intervention (36 PA sessions, 12 vs 20 weeks depending on assignment)
  Change in aerobic fitness

SECONDARY OUTCOMES:
Body composition | At the end of the intervention (36 PA sessions, 12 vs 20 weeks depending on assignment)
  Change in body composition
BMI | At the end of the intervention (36 PA sessions, 12 vs 20 weeks depending on assignment)
  Change in BMI
HbA1c | At the end of the intervention (36 PA sessions, 12 vs 20 weeks depending on assignment)
  Change in HbA1c
Lipid values | At the end of the intervention (36 PA sessions, 12 vs 20 weeks depending on assignment)
  Change in Lipid values
Motor performance | At the end of the intervention (36 PA sessions, 12 vs 20 weeks depending on assignment)
  Change in motor performance
Physical activity | At the end of the intervention (36 PA sessions, 12 vs 20 weeks depending on assignment)
  Change in physical activity
Well-being | At the end of the intervention (36 PA sessions, 12 vs 20 weeks depending on assignment)
  Change in well-being (validated questionnaire)
Self-efficacy | At the end of the intervention (36 PA sessions, 12 vs 20 weeks depending on assignment)
  Change in self-efficacy (questionnaire)
Qualitative evaluation (satisfaction of achievement of personal objectives, evaluation of group session) | At the end of the intervention (36 PA sessions, 12 vs 20 weeks depending on assignment)
Adherence/Attendance: Number of physical activity sessions attended | During the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- University of Lausanne Hospitals, Lausanne, Switzerland

REFERENCES:
- [Derived] Arhab A, Junod N, Rossel JB, Giet O, Sittarame F, Beer S, Sofra D, Durrer D, Delgado H, Castellsague M, Laimer M, Puder JJ. Effectiveness of a real-life program (DIAfit) to promote physical activity in patients with type 2 diabetes: a pragmatic cluster randomized clinical trial. Front Endocrinol (Lausanne). 2023 Jul 3;14:1155217. doi: 10.3389/fendo.2023.1155217. eCollection 2023. PMID 37484961
- [Derived] Allet L, Giet O, Barral J, Junod N, Durrer D, Amati F, Sykiotis GP, Marques-Vidal P, Puder JJ. Educational Level Is Related to Physical Fitness in Patients with Type 2 Diabetes - A Cross-Sectional Study. PLoS One. 2016 Oct 12;11(10):e0164176. doi: 10.1371/journal.pone.0164176. eCollection 2016. PMID 27732627
- See also: Website of the program — http://www.diafit.ch